CLINICAL TRIAL: NCT00002747
Title: RANDOMIZED TRIAL OF NEOADJUVANT CHEMOTHERAPY AND SURGERY +/- RADIOTHERAPY VERSUS SURGEERY +/- RADIOTHERAPY IN OPERABLE SQUAMOUS CELL CARCINOMA OF THE ORAL CAVITY
Brief Title: Surgery and Radiation Therapy With or Without Chemotherapy in Treating Patients With Mouth Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064678; CNR-012309
Record Dates: First submitted 1999-11-01; First posted 2004-06-23 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-05

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Fluorouracil

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Procedure: conventional surgery
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known if surgery plus radiation therapy is more effective with or without chemotherapy for treating mouth cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery and radiation therapy with or without chemotherapy in treating patients with stage II, stage III, or stage IV mouth cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the short- and long-term local control rates, disease-free survival, and overall survival following treatment with neoadjuvant cisplatin plus fluorouracil followed by surgery with or without radiotherapy vs surgery alone with or without radiotherapy in patients with previously untreated stage II-IV squamous cell carcinoma of the oral cavity. II. Assess the prognostic significance of clinical and pathologic responses to neoadjuvant chemotherapy in these patients. III. Compare the short- and long-term toxic effects of these two regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center and nodal status (N0 vs N1-2 vs N3). Patients are randomized to one of two treatment arms. Arm I: Patients receive cisplatin IV on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 2 courses or progressive disease at any time proceed to surgery. Patients undergo resection of the primary tumor site and possible nodal dissection no sooner than 2 weeks after completion of chemotherapy. Patients then undergo radiotherapy over 5-6 weeks no later than 8 weeks after surgery. Arm II: Patients undergo surgery and radiotherapy as in arm I. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then yearly thereafter.

PROJECTED ACCRUAL: A total of 240 patients will be accrued for this study over 9 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Squamous cell carcinoma of the lower oral cavity eligible for resection T2 (greater than 3 cm), T3, or T4, and N0-3 M0 (UICC staging system) No requirement for postsurgical reconstruction that would impede further radiotherapy

PATIENT CHARACTERISTICS: Age: 70 and under Performance status: WHO 0 or 1 Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 2,000/mm3 Platelet count at least 110,000/mm3 Hepatic: Not specified Renal: Creatinine no greater than 1.3 mg/dL Creatinine clearance at least 50 mg/mL BUN no greater than 50 mg/dL Cardiovascular: No cardiopathy Other: No significant internal disease No prior malignancy except basal cell carcinoma of the skin No geographic barrier to treatment

PRIOR CONCURRENT THERAPY: No prior therapy

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 1992-09

CONTACTS AND LOCATIONS:
Overall Officials: R. Molinari, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Istituto Nazionale per lo Studio e la Cura dei Tumori, Milan, Italy